CLINICAL TRIAL: NCT01728012
Title: The Prevalence of Cardiovascular Risk Factors in Patients More Than 10 Years Following Successful Renal Transplant.
Brief Title: Long-term Cardiovascular Risk Following Successful Renal Transplantation
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: REK2010/2926
Record Dates: First submitted 2012-11-08; First posted 2012-11-16 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Renal Transplant
Keywords: Successful transplantation; Long-term observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and urine will be collected along with the clinical observations. Serum, plasma and urine will be frozen for later analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- eGFR >=60ml/min/1.73m2: Patients with an estimated glomerular filtration rate of >=60 ml/min/1.73m2.
- eGFR 45-60ml/min/1.73m2: Patients with estimated glomerular filtration rate >=45 ml/min/1.73m2 and <60ml/min/1.73m2.

SUMMARY:
Mineral metabolism disturbances occur early during the course of chronic kidney disease and eventually affect most patients. For how long such disturbances persist after a successful renal transplantation is mainly unknown. This study will investigate the prevalence of such disturbances in patients more than 10 years following a successful renal transplantation. The patients will be recruited from an existing registry in Norway.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the Norwegian Renal Registry
* Documented elevated iPTH at Tx and 10 weeks post-tx
* Well functioning transplant 10 years following tx
* Signed informed consent

Exclusion Criteria:

* Lack of ability to comply with the protocol
* Refused written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients registered in the Norwegian Renal Registry with transplan more than 10 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Fibroblast growth factor 23 (FGF23) | More than 10 years after successful renal transplantation
  To evaluate the long-term effect of a successful renal transplant on this biomarker.

SECONDARY OUTCOMES:
Intact parathyroid hormone (iPTH) | More than 10 years after successful renal transplantation
  To evaluate the long-term effect of a successful renal transplant on this biomarker.
Klotho | More than 10 years after successful renal transplantation
  To evaluate the long-term effect of a successful renal transplant on this biomarker.
Neutrophil gelatinase-associated lipocalin (NGAL) | More than 10 years after successful renal transplantation
  To evaluate the long-term effect of a successful renal transplant on this biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Hjørdis Bleskestad, MD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway